CLINICAL TRIAL: NCT02160379
Title: Dynamic Effect of Gastrointestinal Hormones on Cerebral Mechanisms Involved in Brain Perception of Food Pictures After Bariatric Surgery
Brief Title: Effects of Roux-en-Y Gastric Bypass on Gastro-intestinal Hormone Secretion and Brain Responses Food Pictures
Status: Completed | Type: Observational
Sponsor: University of Lausanne (Other)
Responsible Party: Principal Investigator, Luc Tappy, MD, Professor of Physiology, University of Lausanne
Other Study IDs: 219/09
Record Dates: First submitted 2014-06-04; First posted 2014-06-10 (Estimated); Last update posted 2014-06-10 (Estimated); Status verified 2014-06

CONDITIONS: Obesity
Keywords: roux-en-Y-gastric bypass; brain responses to food; gastrointestinal hormones; bile acids
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- post Roux-en-Y-gastric bypass: Formerly obese females 1-5 years after gastric bypass
  Interventions: Other: standard test meal
- matched controls: non-operated females age-and weight-matched to post Roux-en-Y-gastric bypass subjects
  Interventions: Other: standard test meal
- healthy young controls: non overweight (BMI between 19 and 25 kg/m2) healthy females
  Interventions: Other: standard test meal

INTERVENTIONS:
Other: standard test meal

SUMMARY:
This is a cross-sectional study enrolling

* 11 weight-stable, formerly obese female patients 1-5 years after Roux-en-Y gastric Bypass (RYGB)
* 11 age- and weight-matched female subjects
* 10 normal weight (Body Mass Index 19-25 kg/m2) subjects The following measurements will be performed in each participants in basal conditions (after an overnight fast) and after ingestion of a standard meal
* electroencephalographic recordings of visually evoked potential after presentation of food- or non-food pictures
* plasma concentration of metabolites (glucose, fatty acids), glucoregulatory hormones (insulin, glucagon), gastro-intestinal hormones (Gastric Inhibitory Polypeptide (GIP), Glucagon-like Peptide-1 (GLP1), ghrelin,Cholecystokinin (CCK), and bile acids Aims of this observational study are
* to evaluate the effects of RYGB on brain perception of food related visual stimulation
* to search for relationships between RYGB effects on brain responses and gastro-intestinal hormone secretion

ELIGIBILITY:
Inclusion Criteria:

* good apparent health
* gender: female
* age 18-50
* non-smoker

Exclusion Criteria:

* diabetes or antidiabetic medication
* consumption of more than 50g alcohol per week
* vegetarian or any special diet

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Formerly obese patients attending the obesity clinics of Lausanne University Hospital and healthy subjects resident in the Lausanne area
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2011-01; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Changes of visually-evoked EEG potentials after ingestion of a meal | basal, 120 min postprandial and 240 postprandial
  Recording and analysis of visual evoked potentials (VEPs) while patients categorize photographs of foods and non-food kitchen utensils

SECONDARY OUTCOMES:
changes in plasma triglyceride concentration after ingestion of a meal | basal, 90 min postprandial and 180 postprandial
  Measurement of triglyceride concentrations at 30-60 min intervals in basal conditions (after an overnight fast) and over 6 hours after ingestion of a standard meal)
Changes in plasma glucoincretins (GLP1 and GIP) concentrations after ingestion of a meal | basal, 90 min postprandial and 180 postprandial
  Measurement of GLP1 and GIP concentrations at 30-60 min intervals in basal conditions (after an overnight fast) and over 6 hours after ingestion of a standard meal)
Changes in plasma cholecystokinin concentrations after ingestion of a meal | basal, 90 min postprandial and 180 postprandial
  Measurement of cholecystokinin concentrations at 30-60 min intervals in basal conditions (after an overnight fast) and over 6 hours after ingestion of a standard meal)
Changes in plasma bile acids concentrations after ingestion of a meal | basal, 90 min postprandial and 180 postprandial
  Measurement of bile acids concentrations at 30-60 min intervals in basal conditions (after an overnight fast) and over 6 hours after ingestion of a standard meal)
changes in plasma glucoregulatory status after ingestion of a meal | basal, 90 min postprandial and 180 postprandial
  Measurement of glucose, insulin, glucagon and non-esterified fatty acid concentrations at 30-60 min intervals in basal conditions (after an overnight fast) and over 6 hours after ingestion of a standard meal)

CONTACTS AND LOCATIONS:
Overall Officials: Luc Tappy, MD, Principal Investigator — University of Lausanne
Locations (1):
- CHUV-clinical research center, Lausanne, Canton of Vaud, Switzerland